CLINICAL TRIAL: NCT05932329
Title: Reducing Free Sugar Intakes: A Role for Sweet Taste II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RFSII2023
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Dietary Behaviour
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: randomized intervention design
Who Masked: Investigator, Outcomes Assessor
Masking Description: All researchers in contact with participants will be blinded, and all analysts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sweet Taste (Active Comparator): The intervention will be provided to participants in written form, in an opaque sealed envelope.
  Interventions: Behavioral: Dietary Advice
- Taste (Active Comparator): The intervention will be provided to participants in written form, in an opaque sealed envelope.
  Interventions: Behavioral: Dietary Advice
- No Taste (Active Comparator): The intervention will be provided to participants in written form, in an opaque sealed envelope.
  Interventions: Behavioral: Dietary Advice

INTERVENTIONS:
Behavioral: Dietary Advice — Dietary Advice provided

SUMMARY:
This randomised controlled trial aims to assess the effects of three different types of dietary advice for reducing free sugar intakes, on intakes of free sugar, in a sample of the UK population.

DETAILED DESCRIPTION:
The primary objective of this randomised controlled trial is to assess the effects of three different types of dietary advice, for reducing total energy intakes (TEI) of free sugars. A total of 150 participants (age 18-65 years) consuming diets >5% total energy intake from dietary free sugars will be recruited from across the Dorset region. All participants will be asked to reduce their free sugar intake to <5% TEI, and to aid with this, they will be encouraged to reduce their intakes of specific foods identified as high in free sugars. Participants will also be advised to replace these foods with other foods dependent on their taste. Participants will be randomised to replace high sugar foods with: 1) foods that are low in sugars, but high in sweet taste; 2) food that are low in sugars, but high in other tastes; and 3) foods that are low in taste. The primary outcome will be changes in free sugar consumption from baseline to endpoint at week 4. Secondary outcomes will include change in: BMI; dietary profiles; sweetness preference; sweetness liking; food choices; low calorie sweetened food intakes and adherence levels at week 4.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-65 years;
2. able to provide consent and complete all study materials;
3. consuming >5% of TEI from free sugars;
4. residing in the South of England, and able to attend Bournemouth University for testing.

Exclusion Criteria:

1. individuals who are pregnant or breastfeeding;
2. underweight (BMI <18.5);
3. have pre-existing clinical conditions such as diabetes mellitus, eating disorders, Crohn's disease and other illness's leading to participants receiving external nutritional advice and dietary restrictions;
4. have pre-existing medical conditions affecting swallow ability, taste and smell perception;
5. currently following a specific dietary programme (e.g.: Slimming World);
6. current smokers or have smoked within 3 months of the study start date.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Free sugar intakes | Baseline to week 4
  Percentage energy intake from free sugars, assessed using diet diaries
Adherence | Baseline to week 4
  Adherence to the recommendations provided, assessed using diet diaries and self-reported adherence

SECONDARY OUTCOMES:
Dietary Intakes | Baseline to week 4
  Nutrient composition and taste of dietary intakes, assessed using diet diaries
Body weight | Baseline to week 4
  Body weight, in kg, assessed using researcher measurements
BMI | Baseline to week 4
  BMI, in kg/m2, assessed using researcher measurements
Waist circumference | Baseline to week 4
  Waist circumference, in cm, assessed using researcher measurements
Body fat percentage | Baseline to week 4
  Body fat percentage, assessed using bioimpedence, as conducted by the researcher measurements
Sweet food preferences | Baseline to week 4
  Preferences for various sweet foods/fluids, assessed using a taste test, where participants sample several sweet and non-sweet foods and rate them for pleasantness on a 100mm Visual Analogue Scale. Higher scores signify stronger preferences
Sweet food perceptions | Baseline to week 4
  Perceptions of the strength of sweet taste for various sweet foods/fluids, assessed using a taste test, where participants sample several sweet and non-sweet foods and rate them for strength of taste on a 100mm Visual Analogue Scale. Higher scores signify stronger perceptions
Sweet food intakes | Baseline to week 4
  Selection of sweet foods/fluids at a given meal, assessed where participants can consume freely from a meal composed of sweet and non-sweet foods, and proportion of sweet foods consumed is measured in terms of weight consumed
Sweet food attitudes | Baseline to week 4
  Attitudes towards sugar, sweeteners, and sweet-tasting foods, assessed using a questionnaire, soon to be published. Higher scores denote stronger attitudes.
Adverse events | Baseline to week 4
  Adverse events, assessed by self-report
Eating-based attitudes | Baseline to week 4
  Attitudes towards eating, assessed using the Three Factor Eating Questionnaire (Karlsson J, et al. IJO 2000; 24: 1715-1725)
Subjective Quality of Life | Baseline to week 4
  Quality of Life, measured using the SF-36 questionnaire (Ware et al, 1996), where Quality of Life is assessed out of 100, where a higher score demonstrates better quality of life
Barriers and facilitators to success | Baseline to week 4
  An assessment of barriers and facilitators to success, assessed by self-report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Appleton, Principal Investigator — Bournemouth University
Locations (1):
- Bournemouth University, Bournemouth, US and Canada Only, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared with other researchers on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From publication of the results

REFERENCES:
- See also: This study is linked to study registration NCT05684757 — https://www.clinicaltrials.gov